CLINICAL TRIAL: NCT03095755
Title: Ischemic Conditioning as an Intervention to Improve Motor Function in Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Marquette University (Other)
Responsible Party: Principal Investigator, Matthew Durand, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO00019103
Record Dates: First submitted 2017-03-23; First posted 2017-03-30 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ischemic Conditioning (Experimental): The investigators will perform ischemic conditioning on the paretic leg by inflating a blood pressure cuff to 225 mmHg to occlude blood flow to the leg for 5 minutes. This will be repeated for 5 cycles, with 5 minutes of rest between each cycle. The intervention will be performed for a maximum of 12 times within a 4 week period.
  Interventions: Other: Ischemic Conditioning
- Sham (Sham Comparator): The investigators will perform sham ischemic conditioning on the paretic leg by inflating a blood pressure cuff to only 25 mmHg on the leg for 5 minutes. This will be repeated for 5 cycles, with 5 minutes of rest between each cycle. The intervention will be performed for a maximum of 12 times within a 4 week period.
  Interventions: Other: Sham

INTERVENTIONS:
Other: Ischemic Conditioning — Inflation of blood pressure cuff to 225 mmHg on paretic leg. 1 session: 5 minutes of inflation, 5 minutes deflation, repeated 5 times. Maximum 12 sessions over 4 weeks.
  Arms: Ischemic Conditioning
Other: Sham — Inflation of blood pressure cuff to 25 mmHg on paretic leg. 1 session: 5 minutes of inflation, 5 minutes deflation, repeated 5 times. Maximum 12 sessions over 4 weeks.
  Arms: Sham

SUMMARY:
The investigators will test whether an intervention called ischemic conditioning can improve paretic leg motor function in chronic stroke subjects.

DETAILED DESCRIPTION:
This study will study ischemic conditioning (IC) as an intervention to improve motor function post-stroke. IC is a well studied, well tolerated intervention which has been shown to improve regional blood flow, motor neuron excitability and muscle function in multiple patient groups and in young, healthy subjects. Because IC targets three physiological systems which are all affected by stroke, the investigators hypothesize that repeated bouts of IC will result in improved motor function of the paretic leg.

ELIGIBILITY:
Inclusion Criteria:

1. be between the ages of 18-85
2. able to give informed consent
3. be ≥ 6 months post diagnosis of unilateral cortical stroke and
4. have residual leg paresis.

Exclusion Criteria:

1. chronic low back or hip pain
2. substance abuse
3. head trauma in last 6 months
4. neurodegenerative disorder
5. any uncontrolled medical condition
6. any condition where knee extension contractions are contraindicated
7. people who are unable to follow multi step commands.
8. people who cannot walk ≥ 10 ft without physical assistance.
9. history of major psychiatric disorder
10. participant has had a myocardial infarction in the last year
11. participant has uncontrolled hypertension
12. participant is unable to contract knee muscles

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Leg Muscle Strength | Within 1 year of admission into the study
  Maximum voluntary contraction of the leg muscles, measured in Newton Meters, as assessed using a Biodex dynamometer.

SECONDARY OUTCOMES:
Leg Muscle Fatigue | Within 1 year of admission into the study
  Duration the leg muscles can sustain contraction to a load level equal to 30% of a maximum voluntary contraction. Measurement units will be seconds the contraction can be held, as assessed using a Biodex Dynamometer.
Brachial Artery Flow Mediated Dilation | Within 1 year of admission into the study
  Percent dilation of the brachial artery

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Durand, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Marquette University, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided